CLINICAL TRIAL: NCT05755425
Title: CPAP Versus High Flow Nasal Cannula Oxygen for the Treatment of Patients With Community Acquired Pneumonia Induced Acute Hypoxemic Respiratory Failure in the Ward
Brief Title: CPAP Versus HFNO for the Treatment of Acute Hypoxemic Respiratory Failure Due to Community Acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Evangelismos Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, IOANNA SIGALA, Pulmonologist-Intensivist, Evangelismos Hospital
Other Study IDs: 139/05-05-2022
Record Dates: First submitted 2023-02-11; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Pneumonia; Respiratory Failure
Keywords: CPAP; HFNO
MeSH Terms: conditions — Pneumonia; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPAP: When a patient needs FiO2 >50% to keep SpO2 >93%, or SpO2 >95% in case of persistent respiratory distress defined as RR>35/min, full face CPAP will be applied
  Interventions: Device: CPAP
- HFNO: When a patient needs FiO2 >50% to keep SpO2 >93%, or SpO2 >95% in case of persistent respiratory distress defined as RR>35/min, HFNO will be applied
  Interventions: Device: HFNO

INTERVENTIONS:
Device: CPAP — CPAP will be delivered with a CPAP valve with venturi flow system with full-face mask. Treatment will start with CPAP set at 10cmH2O and FiO2 60% to target a SpO2 ≥90% or PO2 ≥60mmHg and then adjusted according to SpO2, respiratory distress and clinical tolerance
  Groups: CPAP
Device: HFNO — HFNO will be applied initially at maximal settings: 100% FiO2, flow rate 60 L/min and temperature 37C . Within 1 to 2 h, the HFNO settings should be titrated based on patients respiratory rate (<25-30 per minute), SpO2 (92-96%) and comfort
  Groups: HFNO

SUMMARY:
the study compares two non-invasive respiratory support modalities ie CPAP and High Flow nasal cannula oxygen for the treatment of severe hypoxemic respiratory failure attributed to Community acquired Pneumonia.

DETAILED DESCRIPTION:
CPAP and High Flow nasal cannula oxygen are two established modalities for non-invasive respiratory support . In COVID pandemic era both CPAP and HFNO were widely used in the ward for the treatment of COVID-19 induced acute hypoxemic respiratory failure in order to prevent progression to intubation. Head to head comparison between the two modalities mentioned for the treatment of severe hypoxemic respiratory failure is not available neither in COVID pneumonia or Community acquired pneumonia (CAP).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age >18 year old.
* Been hospitalized with community acquired pneumonia
* hospitalized in common ward (not ICU)
* Patients should have pneumonia- pulmonary infiltrates in chest-xray and hypoxemic respiratory failure.
* Patients should be unable to keep: SpO2>93% with FiO2 50%, or SpO2 95% with FiO2 50% and have evidence of respiratory distress defined as Respiratory rate -RR>35/min

Exclusion Criteria:

* Need for immediate or imminent intubation
* not fit for escalation of treatment: defined as intubation, mechanical ventilation and ICU support.
* Pregnant women
* Contraindication to CPAP or HFNO

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients with community acquired pneumonia induced acute hypoxemic respiratory failure that are hospitalized in the common ward and need FiO2 >50% to keep SpO2 >93%, or SpO2 >95% in case of persistent respiratory distress defined as RR>35/min.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
days free from ventilatory support | 28 days
  days without support with either mechanical ventilation, HFNO, CPAP

SECONDARY OUTCOMES:
treatment failure defined | 28 days
  no of patients that needed intubation and invasive mechanical ventilation or died
intubation rate | 28 days
hospital mortality | 28 days
days under non-invasive respiratory support | 28 days
  days without support with HFNO or CPAP
hospital length of stay | 28 days
Partial pressure of oxygen PaO2 change at 2h, 12h and 24h | 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Evaggelismos Hospital, Athens, Attica
  - University General Hospital of Larissa, Larissa, Thesaly